CLINICAL TRIAL: NCT05196464
Title: ACT Workshops: A Novel Delivery Modality to Increase Access to Care for Rural Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1576467
Record Dates: First submitted 2021-12-14; First posted 2022-01-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Access to Care; Psychological Distress
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: two intervention randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VA primary care patients (Other): VA primary care patients with psychological distress are being enrolled
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) Workshop; Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) Workshop — ACT workshops are single-day workshops that last 5-6 hours. The workshops will 1) Acceptance and Mindfulness Training emphasizing new ways of managing troubling thoughts, feelings, and physical sensations (e.g., learning how to recognize, and develop cognitive distance from unhelpful thoughts) and strategies to willingly face experiences that cannot be changed; and 2) Committed Action Training to help Veterans clarify what matters most to them (e.g., valued domains including family, friends, spirituality, career) and what they want to stand for in life, how they want to behave, and what strengths and qualities they want to develop. Within this context, the workshop will encourage engagement in, rather than avoidance of, actions consistent with valued directions, including engagement in healthcare. Workshop participants will be given homework related to implementing a key coping skill.
Behavioral: Treatment as usual (TAU) — TAU will consist of a consult to a mental health provider at their rural clinic. The patient will then be scheduled for an intake and offered traditional mental health treatment options. Treatment options are likely to include outpatient individual psychotherapy, psychotherapy groups, or medication management.

SUMMARY:
This study investigates access, effectiveness, and acceptability of 1-day ACT workshops on problematic mental health symptoms.

DETAILED DESCRIPTION:
This study proposes to investigate access, effectiveness, and acceptability of 1-day ACT workshops delivered in 2 rural VA primary clinics with 32 Veterans with problematic mental health symptoms (i.e., depression, PTSD, or anxiety) that are risk factors for suicide.

ELIGIBILITY:
Inclusion Criteria:

* 1) current mental health symptoms as measured by one of the following indicators: PHQ-9 ≥ 10, PCL-5 ≥ 30, or GAD-7 ≥ 10.

Exclusion Criteria:

1. cognitive impairment measured by BOMC,
2. current psychosis or mania as evidenced in the medical record,
3. current suicidal intent as measured by the P4,
4. use of mental health services within or outside of VA in the last 6 months as measured by CPRS and the non-VA services questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Access to mental health care | 1 month
  Access to care is measured by hours of active treatment Veterans receive within and outside of VA.
Psychological Distress | 1 month
  Psychological distress as measured by the Depression, Anxiety, and Stress Scale (DASS-21). Score range on 0-42. Higher scores indicate greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse Veterans Affairs Medical Center, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No